CLINICAL TRIAL: NCT05016219
Title: Phase 2 - The Use of Rhythmic Light Therapy to Entrain Gamma Oscillations and the Circadian System in Patients With Alzheimer's Disease
Brief Title: Phase 2 - Rhythmic Light Therapy for Alzheimer's Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Population Health Science and Policy, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 21-0378-02
Record Dates: First submitted 2021-08-12; First posted 2021-08-23 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment
Keywords: Light Treatment; Circadian Rhythms; Gamma Wave Entrainment; Rhythmic Light; Sleep; Cognition
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Intervention plus Active Rhythm (Active Comparator): The device will set on a tabletop in a room where the participant spends at least 2 hours in the morning. Using a timer, it will automatically turn on at preferred wakeup times (but no later than 09:00 am) chosen by the participant. Lights will remain on for at least 2 hours and participants will be asked to remain the space that lights are being applied for that period of time.
  Interventions: Device: Circadian-Effective Light; Device: Rhythmic Light
- Active Light plus Placebo Rhythm (Active Comparator): The device will set on a tabletop in a room where the participant spends at least 2 hours in the morning. Using a timer, it will automatically turn on at preferred wakeup times (but no later than 09:00 am) chosen by the participant. Lights will remain on for at least 2 hours and participants will be asked to remain the space that lights are being applied for that period of time.
  Interventions: Device: Circadian-Effective Light; Device: Placebo Rhythmic Light
- Placebo Light plus Active Rhythm (Active Comparator): The device will set on a tabletop in a room where the participant spends at least 2 hours in the morning. Using a timer, it will automatically turn on at preferred wakeup times (but no later than 09:00 am) chosen by the participant. Lights will remain on for at least 2 hours and participants will be asked to remain the space that lights are being applied for that period of time.
  Interventions: Device: Rhythmic Light; Device: Placebo Light
- Placebo Light plus Placebo Rhythm (Placebo Comparator): The device will set on a tabletop in a room where the participant spends at least 2 hours in the morning. Using a timer, it will automatically turn on at preferred wakeup times (but no later than 09:00 am) chosen by the participant. Lights will remain on for at least 2 hours and participants will be asked to remain the space that lights are being applied for that period of time.
  Interventions: Device: Placebo Light; Device: Placebo Rhythmic Light

INTERVENTIONS:
Device: Circadian-Effective Light — Narrowband blue light
  Other Names: Active Light
  Arms: Active Intervention plus Active Rhythm; Active Light plus Placebo Rhythm
Device: Rhythmic Light — 40 hertz (Hz) flicker
  Arms: Active Intervention plus Active Rhythm; Placebo Light plus Active Rhythm
Device: Placebo Light — Narrowband red light
  Arms: Placebo Light plus Active Rhythm; Placebo Light plus Placebo Rhythm
Device: Placebo Rhythmic Light — Random flicker for placebo rhythmic effect
  Arms: Active Light plus Placebo Rhythm; Placebo Light plus Placebo Rhythm

SUMMARY:
Participants will randomly be placed into one of four groups and experience one of the four following conditions: (1) a placebo light that provides a 40 hertz (Hz) flicker (rhythmic light [RL]); (2) a placebo light with a random flicker (placebo condition for rhythmic light); (3) a light source that will stimulate the circadian system and provides a 40 Hz flicker (RL); or (4) a light source that will stimulate the circadian system and provides a random flicker (placebo condition for rhythmic light). Following a baseline week, participants will experience his/her assigned lighting condition for two hours in the morning for 8 weeks. After a 4-week washout period, a final round of assessments will be obtained. Study assessments (except for the Pittsburgh Sleep Quality Index and Montreal Cognitive Assessment) will be collected at the end of each week, for a total of 8 assessments.

DETAILED DESCRIPTION:
The tailored lighting intervention used to promote circadian entrainment will provide high circadian stimulation during the day produced by narrowband blue light peaking at 470 nanometers (nm). A comparison lighting intervention (i.e., placebo lighting), a narrowband red light peaking at 630 nm, will be used as a control. Both the red and the blue light devices will also provide either the 40 hertz (Hz) flicker (RL) or the random flicker (placebo RL). For the random flicker (placebo RL), the duty cycle will be delivered with a random interval determined by a Poisson process with an average interval of 40 hertz (Hz).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with mild cognitive impairment or mild Alzheimer's disease, as defined by a Montreal Cognitive Assessment score between 17 and 25;
* Have sleep disturbance indicated by a score >5 on the Pittsburgh Sleep Quality Index
* Participants must reside in their homes, independent living, or assisted living facilities

Exclusion Criteria:

* Participants taking sleep medication
* Residence in a skilled nursing facility or long-term care
* Obstructing cataracts, macular degeneration, and blindness
* Severe sleep apnea or restless leg syndrome
* History of severe epilepsy

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Cognition using the Montreal Cognitive Assessment (MoCA) | baseline
  The Montreal Cognitive Assessment is a one-page, 30-point test that can be administered in 10 minutes. It assesses short-term memory, visuospatial abilities, executive functions, attention, concentration and working memory, language, and orientation to time and place. total score ranging from 0 to 30 units on a scale, with higher score indicating better cognitive global function.
Cognition using the Montreal Cognitive Assessment (MoCA) | at the end of week 9
  The Montreal Cognitive Assessment is a one-page, 30-point test that can be administered in 10 minutes. It assesses short-term memory, visuospatial abilities, executive functions, attention, concentration and working memory, language, and orientation to time and place. total score ranging from 0 to 30 units on a scale, with higher score indicating better cognitive global function.
Cognition using the Montreal Cognitive Assessment (MoCA) | at the end of week 14
  The Montreal Cognitive Assessment is a one-page, 30-point test that can be administered in 10 minutes. It assesses short-term memory, visuospatial abilities, executive functions, attention, concentration and working memory, language, and orientation to time and place. total score ranging from 0 to 30 units on a scale, with higher score indicating better cognitive global function.

SECONDARY OUTCOMES:
Cognition using a working memory task | baseline
  Participants view a serial visual display of letters and math problems. They are asked to hold the letters in memory while simultaneously determining if the simple math problems are correct (e.g., 7+5=13). Math performance is measured in percent correct and verbal performance is assessed by calculating Accuracy and Reaction Time (RT).
Cognition using a working memory task | at the end of week 9
  Participants view a serial visual display of letters and math problems. They are asked to hold the letters in memory while simultaneously determining if the simple math problems are correct (e.g., 7+5=13). Math performance is measured in percent correct and verbal performance is assessed by calculating Accuracy and Reaction Time (RT).
Cognition using a working memory task | at the end of week 14
  Participants view a serial visual display of letters and math problems. They are asked to hold the letters in memory while simultaneously determining if the simple math problems are correct (e.g., 7+5=13). Math performance is measured in percent correct and verbal performance is assessed by calculating Accuracy and Reaction Time (RT).
Cognition using a word pair associates task | baseline
  Participants are presented with 48 word-pairs in the evening. Recognition tests are assessed both immediately following the encoding session, and delayed during retrieval.
Cognition using a word pair associates task | at the end of week 9
  Participants are presented with 48 word-pairs in the evening. Recognition tests are assessed both immediately following the encoding session, and delayed during retrieval.
Cognition using a word pair associates task | at the end of week 14.
  Participants are presented with 48 word-pairs in the evening. Recognition tests are assessed both immediately following the encoding session, and delayed during retrieval.
Cognition using an implicit priming task | baseline
  Participants will be presented with simple pictures of objects and animals. Following a break, the participant will then be asked to identify a larger set of pictures as soon as he/she is able to do so as the pictures clarify over time; some of these test pictures were shown previously and some are new.
Cognition using an implicit priming task | at the end of week 9
  Participants will be presented with simple pictures of objects and animals. Following a break, the participant will then be asked to identify a larger set of pictures as soon as he/she is able to do so as the pictures clarify over time; some of these test pictures were shown previously and some are new.
Cognition using an implicit priming task | at the end of week 14.
  Participants will be presented with simple pictures of objects and animals. Following a break, the participant will then be asked to identify a larger set of pictures as soon as he/she is able to do so as the pictures clarify over time; some of these test pictures were shown previously and some are new.
Cognition using the Alzheimer's Disease Assessment Scale - Cognitive Subscale | baseline
  This interview-style test assesses multiple cognitive domains such as memory, language, praxis, and orientation. The ADAS-Cog subscale is scored from 0-100. The full ADAS is scored from 0 to 150 by summing the number of errors made on each task so that higher scores indicate worse performance.
Cognition using the Alzheimer's Disease Assessment Scale - Cognitive Subscale | at the end of week 9
  This interview-style test assesses multiple cognitive domains such as memory, language, praxis, and orientation. The Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) subscale is scored from 0-100. The full ADAS is scored from 0 to 150 by summing the number of errors made on each task so that higher scores indicate worse performance.
Cognition using the Alzheimer's Disease Assessment Scale - Cognitive Subscale | at the end of week 14.
  This interview-style test assesses multiple cognitive domains such as memory, language, praxis, and orientation. The ADAS-Cog subscale is scored from 0-100. The full ADAS is scored from 0 to 150 by summing the number of errors made on each task so that higher scores indicate worse performance.
Urine Melatonin Biomarker | baseline
  Urine Melatonin Biomarker via urine collection
Urine Melatonin Biomarker | at the end of week 9.
  Urine Melatonin Biomarker via urine collection
Light Exposure using a Daysimeter | baseline
  The Daysimeter will also be used to monitor the total amount of circadian light received by the participant during the study.
Light Exposure using a Daysimeter | week 9
  The Daysimeter will also be used to monitor the total amount of circadian light received by the participant during the study.
Light Exposure using a Daysimeter | week 14.
  The Daysimeter will also be used to monitor the total amount of circadian light received by the participant during the study.
Sleep Quantity using Actigraphy | baseline
  Sleep Quantity measured using Actigraphy
Sleep Quantity using Actigraphy | week 9
  Sleep Quantity measured using Actigraphy
Sleep Quantity using Actigraphy | week 14
  Sleep Quantity measured using Actigraphy
Sleep Quality using the Pittsburgh Sleep Quality Index (PSQI) | baseline
  The Pittsburgh Sleep Quality Index is a tool that can be used to measure sleep quality in clinical populations, composed of 19 items that generate 7 component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction). Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, with higher score indicates worse sleep quality
Sleep Quality using the Pittsburgh Sleep Quality Index (PSQI) | at the end of week 9
  The Pittsburgh Sleep Quality Index is a tool that can be used to measure sleep quality in clinical populations, composed of 19 items that generate 7 component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction). Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, with higher score indicates worse sleep quality
Sleep Quality using the Pittsburgh Sleep Quality Index (PSQI) | at the end of week 14.
  The Pittsburgh Sleep Quality Index is a tool that can be used to measure sleep quality in clinical populations, composed of 19 items that generate 7 component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction). Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, with higher score indicates worse sleep quality
Quality of Life using the Dementia Quality of Life Instrument | baseline
  The Dementia Quality of Life Instrument (DQoL) measures self-esteem, positive affect/humor, negative affect, feelings of belonging, and sense of aesthetics.The DQoL consists of 29 items, grouped into 5 subscales according to domain. Subjects are instructed to answer using a 5-point response scale (score from 1-5), either verbally or through use of a visual scale. Scores for each subscale are Self-esteem (4-20), Positive Affect/Humor (6-30), Absence of Negative Affect (11-55), Feelings of Belonging (3-15), Sense of Aesthetics (5-25); however, subscale scores are not summed for a total score. A higher number indicates greater quality of life.
Quality of Life using the Dementia Quality of Life Instrument | at the end of week 9
  The Dementia Quality of Life Instrument (DQoL) measures self-esteem, positive affect/humor, negative affect, feelings of belonging, and sense of aesthetics.The DQoL consists of 29 items, grouped into 5 subscales according to domain. Subjects are instructed to answer using a 5-point response scale (score from 1-5), either verbally or through use of a visual scale. Scores for each subscale are Self-esteem (4-20), Positive Affect/Humor (6-30), Absence of Negative Affect (11-55), Feelings of Belonging (3-15), Sense of Aesthetics (5-25); however, subscale scores are not summed for a total score. A higher number indicates greater quality of life.
Quality of Life using the Dementia Quality of Life Instrument | at the end of week 14.
  The Dementia Quality of Life Instrument (DQoL) measures self-esteem, positive affect/humor, negative affect, feelings of belonging, and sense of aesthetics.The DQoL consists of 29 items, grouped into 5 subscales according to domain. Subjects are instructed to answer using a 5-point response scale (score from 1-5), either verbally or through use of a visual scale. Scores for each subscale are Self-esteem (4-20), Positive Affect/Humor (6-30), Absence of Negative Affect (11-55), Feelings of Belonging (3-15), Sense of Aesthetics (5-25); however, subscale scores are not summed for a total score. A higher number indicates greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Figueiro, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Light and Health Research Center, Menands, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Background] Rea MS, Figueiro MG, Bullough JD, Bierman A. A model of phototransduction by the human circadian system. Brain Res Brain Res Rev. 2005 Dec 15;50(2):213-28. doi: 10.1016/j.brainresrev.2005.07.002. Epub 2005 Oct 7. PMID 16216333
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Rosen WG, Mohs RC, Davis KL. A new rating scale for Alzheimer's disease. Am J Psychiatry. 1984 Nov;141(11):1356-64. doi: 10.1176/ajp.141.11.1356. PMID 6496779
- [Background] Figueiro MG, Hamner R, Bierman A, Rea MS. Comparisons of three practical field devices used to measure personal light exposures and activity levels. Light Res Technol. 2013 Aug;45(4):421-434. doi: 10.1177/1477153512450453. PMID 24443644
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Hoch CC, Yeager AL, Kupfer DJ. Quantification of subjective sleep quality in healthy elderly men and women using the Pittsburgh Sleep Quality Index (PSQI). Sleep. 1991 Aug;14(4):331-8. PMID 1947597
- [Background] Hughes CP, Berg L, Danziger WL, Coben LA, Martin RL. A new clinical scale for the staging of dementia. Br J Psychiatry. 1982 Jun;140:566-72. doi: 10.1192/bjp.140.6.566. PMID 7104545
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] McKhann G, Drachman D, Folstein M, Katzman R, Price D, Stadlan EM. Clinical diagnosis of Alzheimer's disease: report of the NINCDS-ADRDA Work Group under the auspices of Department of Health and Human Services Task Force on Alzheimer's Disease. Neurology. 1984 Jul;34(7):939-44. doi: 10.1212/wnl.34.7.939. PMID 6610841